CLINICAL TRIAL: NCT02124343
Title: A Pilot Study to Examine the Effect of Acute Exercise on Neutrophil Function in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Exercise and Neutrophil Function in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hywel Dda Health Board (Other)
Responsible Party: Principal Investigator, Alex Jenkins, Research Student, Hywel Dda Health Board
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14/WA/0022
Record Dates: First submitted 2014-04-07; First posted 2014-04-28 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Airway Disease; Neutrophil Function Disorder
Keywords: Neutrophil; Exercise; COPD; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interval Exercise (Experimental): Subjects will undertake an interval exercise session (on a harnessed treadmill) (HP Cosmos Mercury 4.0, HP Cosmos Sports and Medical Gmbh, Nussdorf-Traustein,Germany) based on the average speed calculated from the 6 minute walk test (6MWT).
  Intervals are based on the work previously done by Mador et al., 2009 who used intervals of 150% (for 1 minute) followed by intervals of 75% (for 2 minutes) based on 80% average speed from the 6 minute walk test.
  This study repeated these intervals 7 times with a duration of 23 minutes in total for the exercise intervention with the 75% intervals at the start and at the end of the exercise session. No warm up was undertaken for this method as it was a walking exercise test and the risk of injury was minimised with use of the harnessed treadmill.
  Interventions: Other: Interval Exercise

INTERVENTIONS:
Other: Interval Exercise

SUMMARY:
Exercise is a cornerstone of pulmonary rehabilitation in the treatment of Chronic Obstructive Pulmonary Disease (COPD). Although researchers have shown numerous benefits with exercise in COPD patients, most studies have only looked at exercise tolerance and psychological outcomes following training. COPD is characterised by persistent inflammation that can cause progressive decline in lung function and multisystemic complications. This inflammation can be amplified in patients when they suffer acute exacerbations. There is a wellknown relationship between exercise, immune function and risk of infection. Exercise has also been shown to have an antiinflammatory effect when performed regularly. There is a lack of research looking into the inflammatory or immune response to exercise in patients with COPD. The exercise within this study will be individually tailored to patients with COPD based on their validated 6 minute walk test (6MWT) but the protocol will involve interval exercise that has been used previously. This type of exercise is considered most appropriate for research into mechanisms of benefit because it maintains the exercise training effects of other modalities (e.g. continuous low intensity aerobic exercise) while avoiding the occurrence of limitations to exercise in people with lung problems (e.g. dynamic hyperinflation). It also closely mirrors daily activity of someone with COPD.

The investigators want to explore the effects of exercise specifically on immune function in 15 people COPD and compare any changes to 15 Controls. By better understanding the mechanisms of how exercise affects inflammation, the investigators could eventually design better Pulmonary Rehabilitation interventions, especially for those most at risk.

ELIGIBILITY:
Inclusion Criteria:

* COPD group - 15 Participants who have been diagnosed with any severity of COPD (according to BTS criteria, i.e. >10 pack-year smoking history and post-bronchodilator spirometry FEV1/FVC ratio <0.70 and FEV<80%) and have completed at least 12 from 18 sessions of a pulmonary rehabilitation programme.
* Age 50-80 years.
* Current non-smoker.
* Control group - 15 Participants who will act as Controls, without COPD or cardiovascular disease
* Age 50-80 years (ideally of similar gender distribution)
* Current non-smoker.
* Spirometry: FEV1/FVC>0.7 and FEV>80% predicted

Exclusion Criteria:

* Known asthma or allergic rhinitis or other respiratory disease (bronchiectasis, pulmonary fibrosis).
* A change in any medications within 4 weeks or during the study.
* Require domiciliary oxygen.
* Acute exacerbation of COPD within 4 weeks of study entry.
* Any infection or illness within 4 weeks of study entry.
* Other active inflammatory conditions e.g. rheumatoid arthritis, cancer, unstable cardiac conditions.
* Receiving oral steroids or other immunomodulating drugs.
* Currently undergoing exercise training (including Pulmonary Rehabilitation).
* Any previous cardiovascular contraindications to exercise (e.g. unstable angina).
* Inability to complete the 6MWT due to physical or mental impairment.
* Exhaled CO>10ppm or smoked any cigarettes within 6 months.
* Inability or unwillingness to sign informed consent.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Neutrophil response to exercise | 4 months
  The primary outcome measure for this study is to examine neutrophil responses to acute exercise, including changes in the counts and function of these cells in blood and sputa in order to compare any changes between COPD and age-gender matched controls.

SECONDARY OUTCOMES:
Different health status and the responses on neutrophil function | 4 months
  The secondary outcome measures for this study is to examine the responses of inflammatory (pro and anti) mediators (e.g. cytokines) to acute exercise.

OTHER OUTCOMES:
Effect of inhaled steroids on neutrophil response following exercise | 4 months
  The third outcome for this study is to compare neutrophil response to exercise in those taking different types of inhaled steroid (fluticasone versus budesonide or beclamethasone).
Neutrophil response to exercise in past smokers versus non-smokers | 4 months
  The fourth outcome measure of this study is to compare neutrophil response to exercise in past smokers versus non-smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Jenkins, BSc (Hons), Principal Investigator — Aberystwyth University; Keir E Lewis, MD, Study Chair — Hywel Dda Health Board
Locations (1):
- Prince Philip Hospital, Llanelli, Carmarthenshire, United Kingdom